CLINICAL TRIAL: NCT05646888
Title: Inflammation, Platelets and Sickle Cell Disease
Acronym: Il-Padre
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0255
Record Dates: First submitted 2022-09-06; First posted 2022-12-12 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Platelet Activation; Thromboinflammation; Sickle Cell Disease
Keywords: Sickle cell disease; vaso-occlusive crisis; platelets; thrombo-inflammation
MeSH Terms: conditions — Thromboinflammation; Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Blood sampling — the blood sample will be taken during a planned blood sampling

SUMMARY:
Sickle cell disease (SCD) is an autosomal recessive genetic disorder linked to a single mutation on beta-globin chains. This leads to red blood cell deformation and chronic hemolysis which can result in vaso-occlusive events, anemia and vasculopathy. Pathophysiology is incompletely understood, and beyond red blood cell's abnormalities this involves hemostasis and innate immunity. The aim of our study is to describe the mechanisms of thrombo-inflammation during the vaso-occlusive crisis (VOC) in adults with sickle cell disease.

DETAILED DESCRIPTION:
Pathophysiology of sickle cell disease is incompletely understood. The typical change of red blood cells into sickle cells lead to post-capillary stream abnormalities. This phenomenon is responsible of ischemia-reperfusion injuries. Chronic hemolysis is the second part of the pathophysiology. The consequences are vasoconstriction, endothelial lesions, chronic inflammation, hemostasis and platelets activation. Thrombo-inflammation concept was proposed by Tanguay to describe the interactions between hemostasis, platelets and innate immune cells (neutrophils polynuclear) during thrombotic process. Since this time, this concept was largely described in many clinical situations such as septicemia, COVID-19, coronaropathy, auto-immune diseases and sickle cell disease.

In this project, we will study platelets activation and thrombo-inflammation markers in the beginning of a vaso-occlusive crisis, during the crisis and two months after the crisis. Blood samples will be collected during a routine care sample.

Biological markers studied will be:

* Soluble and surface markers of platelet activation; platelet-leukocytes aggregates
* Plasmatic eicosanoids produced by platelets (TXB2) and immune cells
* In vitro platelets reactivity; dynamic thrombus formation in normal and pathologic arterial blood stream
* Platelet's inflammasome

ELIGIBILITY:
Inclusion Criteria:

* Patient with sickle cell disease diagnosis, hospitalized in emergency department and/or internal medicine department
* Patient older than 18 years
* Written consent to participate to the study
* Patient with health insurance
* Patient able to receive information about the study

Exclusion Criteria:

* Age < 18 years
* Non consent to participate to the study
* Women in pregnancy or breastfeeding
* Treatment with aspirin or non steroidal anti inflammatory drug
* Protected patient
* Patient already involved in a study requiring collection of additional biological samples

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sickle cell disease diagnosis
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate mechanisms of platelet activation in the thrombo-inflammation process during a vaso-occlusive crisis. | First 48h of hospitalization
  by flow cytometry analysis
To evaluate mechanisms of platelet activation in the thrombo-inflammation process during a vaso-occlusive crisis. | Day 13 (+/- 2 days)
  by flow cytometry analysis
To evaluate mechanisms of platelet activation in the thrombo-inflammation process during a vaso-occlusive crisis. | At day 60 (+/- 2 days)
  by flow cytometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Cougoul, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- IUCT-Oncopole University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No